CLINICAL TRIAL: NCT05597683
Title: Quadratus Lumborum Block for Analgesia After Cytoreductive Surgery and Hyperthermic Intra-peritoneal Chemotherapy (CRS and HIPEC): a Double-blind Randomized Controlled Trial
Brief Title: Quadratus Lumborum Block After Cytoreductive Surgery and Hyperthermic Intra-peritoneal Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Young Song, Associate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3-2022-0328
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Cytoreductive Surgery; Hyperthermic Intra-peritoneal Chemotherapy; Peritoneal Cancer

STUDY DESIGN:
Intervention Model Description: hyperthermic intra-peritoneal chemotherapy
Who Masked: Participant, Care Provider
Masking Description: Patients, medical staff who measure outcome variables, and nurses in the recovery room are double-blinded so that medical staff and patients do not know the patient's assigned group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL block group (Experimental): Bilateral transmuscular QL block will be performed under ultrasound-guidance. Twenty mililiter of 0.375% ropivacaine will be injected to each side.
  Interventions: Procedure: Arm I (QL block and multimodal analgesia), Arm II (multimodal analgesia without regional block)
- Control group (No Intervention): QL block will be not performed.

INTERVENTIONS:
Procedure: Arm I (QL block and multimodal analgesia), Arm II (multimodal analgesia without regional block) — Arm I (QL block and multimodal analgesia): Bilateral transmuscular QL block will be done. Postoperative multimodal analgesia including administration of acetaminophen, NSAIDs,nefopam, and rescue opioids
  Arm II (multimodal analgesia without regional block): No block will be done. Postoperative multimodal analgesia including administration of acetaminophen, NSAIDs, nefopam, and rescue opioids
  Arms: QL block group

SUMMARY:
This study aims to assess whether transmusculr quadratus lomborum block (QL block) can reduce postoperative pain after cytoreductive surgery and hyperthermic intra-peritoneal chemotherapy (CRS and HIPEC). Patients will be randomly assigned to either QL block group or control group. Ultrasound-guided bilateral transmuscular quadratus lomborum block will be performed in QL block group using 0.375% ropivacaine. Multimodal analgesic regimen including acetaminophen, nonsteroidal antiinflammatory drugs (NSAIDs), and rescue opioids will be used in every patient. Primary outcome is opioid consumption for 24 hours after surgery. Secondary outcomes included pain scores, time to first rescue analgesics, quality of recovery score, length of hospital stay.

DETAILED DESCRIPTION:
Adult patients scheduled to undergo cytoreductive surgery and hyperthermic intra-peritoneal chemotherapy will be screened for eligibility. After induction of general anesthesia, ultrasound-guided bilateral transmuscular quadratus lomborum block will be done in QL block group. 0.375% ropivacaine will be injected to each side. Patients in control group will receive no block. Multimodal analgesia will be applied to every patient for postoperative pain control. Multimodal analgesic regimen included scheduled administration of acetaminophen, NSAIDs, and rescue opioids. Blinded investigator will assess pain scores at rest and on movement at 6, 12, 24, 48, 72 hours after surgery, analgesic consumptions, nausea, vomiting, and quality of recovery questionnaire.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients who are scheduled to undergo cytoreductive surgery and hyperthermic intra-peritoneal chemotherapy (CRS and HIPEC)

Exclusion Criteria:

1. Allergy to local anesthetics or fentanyl
2. Chronic pain
3. Drug abuse
4. Patients who are unable to use patient-controlled analgesia
5. Skin infection at site for quadratus lomborum block
6. pregnant or breatfeeding women
7. Patients who are unable to communicate

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption for 24 postoperative hours | 24 hours postoperatively
  Total opioid analgesic use for 24 hours after surgery (morphine milligram equivalents (MME))

SECONDARY OUTCOMES:
Analgesic consumption | at postoperative 6, 12, 48, 72 hours
  Analgesic consumption at postoperative 6, 12, 48, 72 hours
Resting pain numeric rating scale(NRS) | at postoperative 6, 12, 24, 48, 72 hours
  Resting pain numeric rating scale(NRS) at postoperative 6, 12, 24, 48, 72 hours.
Numeric rating scale of pain during movement | at postoperative 6, 12, 24, 48, 72 hours
  Numeric rating scale of pain during movement at postoperative 6, 12, 24, 48, 72 hours
Time to first rescue analgesics | within post-operative 24 hours
  Time to first rescue analgesics
Rescue analgesics administration | within post-operative 48 hours
  Rescue analgesics administration count
The incidence of post-operative nausea and vomiting | within post-operative 72 hours
  The incidence of post-operative nausea and vomiting
Patient satisfaction with pain control | At post-operative 72 hours
  Patient satisfaction with pain control in 11 point scale (0-10), The higher the score, the higher the patient's satisfaction
Quality of Recovery Questionnaire (15-item Quality of Recovery) | At post-operative 72 hours
  Each item uses an 11-point numeric rating scale. The sum of the scores of the 15 items ranges from 0 to 150, with a high score indicating good quality of recovery.
Pattern of injectate spread on ultrasonography | During quadratus lumborum (QL) block procedure
  Pattern of injectate spread on ultrasonography
Numeric rating scale at post anesthetic care unit (PACU) | 30 minutes after the end of operation
  Numeric rating scale at post anesthetic care unit. Numeric rating scare is 11-point scale from 0 to 10. The higher the number, the more severe the pain (0 is no pain at all, 10 is the most severe pain imaginable).
Time to first ambulation | within post-operative 72 hours
  Time to first ambulation
Length of hospital stay | within postoperative 30 days
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Young Song, Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No